CLINICAL TRIAL: NCT05967845
Title: Platelet Rich Fibrin Augmented Tympanoplasty Versus Cartilage Tympanoplasty: a Randomized Clinical Trial
Brief Title: Platelet Rich Fibrin Augmented Tympanoplasty Versus Cartilage Tympanoplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Hisham Ebada, Assistant Professor, Mansoura University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: MS.19.04.576
Record Dates: First submitted 2023-06-29; First posted 2023-08-01 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Chronic Suppurative Otitis Media

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Platelet rich fibrin augmented tympanoplasty (Active Comparator): Platelet rich fibrin will be prepaired from the patient's own blood throud a centrifugation process and will be applied on the temproalis fascia graft to improve healing.
  Interventions: Procedure: platelet rich fibrin augmented tympanoplasty
- cartilage tympanoplasty (Active Comparator): A piece of cartilage will be harvested from the concha and used as a graft for tympanoplasty
  Interventions: Procedure: cartilage tympanoplasty

INTERVENTIONS:
Procedure: cartilage tympanoplasty — cartilage tympanoplasty procedure entails repairing the tympanic membrane perforation by using a piece of cartilage harvested from the patient's auricle.
  Arms: cartilage tympanoplasty
Procedure: platelet rich fibrin augmented tympanoplasty — platelet rich fibrin augmented tympanoplasty entails performing the traditional tympanoplasty using the tempralis fascia as a grafting material. However, platelet rich fibrin clot is obtained from the patient's own blood, and applied to the graft to enhance healing process.
  Arms: Platelet rich fibrin augmented tympanoplasty

SUMMARY:
This study was performed to compare healing and hearing outcomes of two tympanoplasty techniques, performed for patients with total or subtotal tympanic membrane perforations. The first group underwent temporalis fascia tympanoplasty, augmented with platelet rich fibrin, while the second group underwent cartilage tympanoplasty. preoperative data, operative techniques, and postoperative outcomes were analyzed.

DETAILED DESCRIPTION:
Two groups are included. In the platelet rich fibrin augmented tympanoplasty group, a piece of temporalis fascia is harvested and used as a graft material. A layer of platelet rich fibrin is added to improve healing process. In the cartilage tympanoplasty group, a piece of cartilage is harvested from the patient concha and used for grafting. Both groups will be compared in terms of healing and hearing. Healing is considered successful if an intact tympanic membrane is achieved withing 12 weeks follow up period. Hearing outcomes are analyzed by comparing the preoperative pure tone audiometry values with the postoperative values.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients older than 18 years.
* Chronic suppurative otitis media mucosal type with total or subtotal perforation.
* Inactive for 3 months.

Exclusion Criteria:

* Recurrent perforation after previous tympanoplasty.
* Active inflammation of middle ear.
* Chronic suppurative otitis media epithelial type.
* Ossicular disruption or fixation diagnosed intraoperatively.
* Immunocompromised patients including uncontrolled diabetics, chronic liver and kidney diseases.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 156 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Healing rate, or graft take rate. | 12 weeks
  Closure of the tympanic membrane perforation. An intact tympanic membrane without residual perforation is considered as adequate healing and successful outcome.

SECONDARY OUTCOMES:
Hearing outcomes | 12 weeks
  Postoperative changes of hearing levels as assessed by pure tone audiometry.

CONTACTS AND LOCATIONS:
Overall Officials: Hisham A Ebada, MD, Principal Investigator — Mansoura University
Locations (1):
- Mansoura University faculty of Medicine, Al Mansurah, Dakahlia Governorate, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Venkatesan D, Umamaheswaran P, Vellikkannu R, Kannan S, Sivaraman A, Ramamurthy S. A Comparative Study of Temporalis Fascia Graft and Full Thickness Tragal Island Cartilage Graft in Type 1 Tympanoplasty. Indian J Otolaryngol Head Neck Surg. 2022 Aug;74(Suppl 1):619-623. doi: 10.1007/s12070-021-02459-2. Epub 2021 Feb 19. PMID 36032890
- [Result] Jain A, Samdani S, Sharma MP, Meena V. Island cartilage vs temporalis fascia in type 1 tympanoplasty: A prospective study. Acta Otorrinolaringol Esp (Engl Ed). 2018 Nov-Dec;69(6):311-317. doi: 10.1016/j.otorri.2017.10.004. Epub 2018 Mar 22. English, Spanish. PMID 29576202
- [Result] Gokce Kutuk S, Ozdas T. Impact of platelet-rich fibrin therapy in tympanoplasty type 1 surgery on graft survival and frequency-specific hearing outcomes: a retrospective analysis in patients with tympanic membrane perforation due to chronic otitis media. J Laryngol Otol. 2019 Dec;133(12):1068-1073. doi: 10.1017/S0022215119002391. Epub 2019 Nov 18. PMID 31735178